CLINICAL TRIAL: NCT06595771
Title: The Incidence of Fibromyalgia in Patients with OUAS and the Effect of CPAP Treatment on Fibromiyalgia Symptom Severity
Brief Title: Obstructive Sleep Apnea Syndrome and Fibromiyalgia
Status: Completed | Type: Observational
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Duygu Geler Külcü, Prof Dr, Haydarpasa Numune Training and Research Hospital
Other Study IDs: FSMEAH-KAEK 2018/37
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2018-08

CONDITIONS: Fibromyalgia, Primary
Keywords: obstructive sleep apnea
MeSH Terms: conditions — Fibromyalgia; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure; Polysomnography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 225 patients with obstructive sleep apnea syndrome: Patients with obstructive sleep apnea syndrome recieved CPAP therapy
  Interventions: Device: continuous positive airway pressure; Device: Polysomnography

INTERVENTIONS:
Device: continuous positive airway pressure — continuous positive airway pressure is a form of positive airway pressure ventilator, which applies mild air pressure on a continuous basis to keep the airways continuously open in people who are able to breathe spontaneously on their own, but need help keeping their airway unobstructed
Device: Polysomnography — Polysomnography measures Apnea-hypopnea index (Minutes)
  Classify and identify Obstructive Sleep Apnea Syndrome (OSAS):
  1. Apnea-hypopnea index: 5-14.9 olan; mild OSAS
  2. Apnea-hypopnea index: 15-29.9: moderate OSAS
  3. Apnea-hypopnea index ≥30: severe OSAS measures duration and percentage of time oxygen saturation dropped below 90% the total minutes of sleep

SUMMARY:
-------------Obstructive sleep apnea syndrome (OSAS) is a syndrome characterized by recurrent complete (apnea) or partial (hypopnea) upper respiratory tract obstruction episodes during sleep and a decrease in blood oxygen saturation. It has been suggested that nocturnal arterial desaturation in patients with OSAS is effective on pain. Intermittent hypoxia and oxidative stress occur in patients with OSAS. Intermittent hypoxia occurring in patients with OSAS causes increased levels of HIF-1-α and mitochondrial reactive oxygen products, resulting in the formation, processing, and formation of central and peripheral synthesis. When the literature is examined, pressure-related pain threshold was measured with algometer in female patients diagnosed with sleep apnea and in the control group, and it was found lower in patients with OSAS.

Fibromyalgia Syndrome (FMS) is a clinical picture with many symptoms such as chronic widespread pain, fatigue, sleep disturbance, cognitive dysfunction. Similar sleep patterns were observed in FMS and OSAS.

In addition to sleep symptoms such as the presence of a similar sleep pattern, a feeling of rest and daytime sleepiness in cases of OSAS and FMS, it has been suggested that these two diseases may be related to each other. Studies examining the relationship between OSAS and FMS syndrome, including sleep disturbance and pain symptoms, are rare in the literature. In the current literature, there are various limitations such as insufficient number of cases, significant difference between demographic characteristics such as gender, ethnicity, age.

Therefore, primary goal of this study is to investigate the association of FMS in patients diagnosed with OSAS. The secondary aim is to investigate the effect of CPAP (Continuous Positive Airway Pressure) treatment on pain sensitivity and symptom severity, functional level, depression in patients diagnosed with FMS, and to investigate the relationship between these parameters and polysomnographic data

DETAILED DESCRIPTION:
Patients between 30-65 years of age who were diagnosed with OSAS according to American Academy of Sleep Medicine (AASM) criteria and who had clinical symptoms of OSAS for at least 1 year before diagnosis will be performed. All OSAS patients recommended and not recommended for CPAP treatment in the sleep clinic will be evaluated according to the American Rheumatology Association (ACR) 1990 and 2016 criteria for FMS. Patients meeting both criteria will be accepted as FMS.

Demographic data and polysomnographic data of patients such as age, height, weight, BMI, occupation, educational status (polysomnographic data (AHI, min. O₂ sat, O₂ saturation <90% elapsed time and percentage, sleep latency, sleep efficacy, REM, nREM1,2,3 polysomnographic data such as times, REM latency, severity of OSAS) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 1-30-65
* Being diagnosed with Obstructive Sleep apnea syndrome and/or having CPAP treatment indication

Exclusion Criteria:

* Chronic inflammatory or autoimmune disease
* hyperthyroidism/hyperthyroidism
* Cognitive dysfunction (such as dementia)
* Severe psychiatric disorder
* Antidepressant medication used in the last 2 weeks
* Non-steroid inflammatory drug used in the last 24 hours

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 30-65 years of age who were diagnosed with OSAS according to American Academy of Sleep Medicine (AASM) criteria and who had clinical symptoms of OSAS for at least 1 year before diagnosis will be performed. All OSAS patients recommended and not recommended for CPAP treatment in the sleep clinic will be evaluated according to the American Rheumatology Association (ACR) 1990 and 2016 criteria for FMS. Patients meeting both criteria will be accepted as FMS.
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Visual Analoge Scale | From enrollment to the end of treatment at 12 weeks
  Mnimum-maximum values: 0-10 Higher scores mean worse outcome for pain scores
Algometer | From enrollment to the end of treatment at 12 weeks
  pain pressure treshold measurements unit: kg/m2 Higher scores mean better outcome
Fibromiyalgia Fatigue Scale Questionnaire | From enrollment to the end of treatment at 12 weeks
  min-max scores:0-72 measures disability Higher scores mean worse outcome
Fibromiyalgia Impact Questionnaire | From enrollment to the end of treatment at 12 weeks"
  measures disability level of patients with Fibromyalgia min-max scores: 0-100 Higher scores mean worse outcome

SECONDARY OUTCOMES:
Epworth Sleepness Scale Questionnaire | From enrollment to the end of treatment at 12 weeks
  measures sleep quality min-max scores: 0-24 score between 16-24 on this scale is considered increased daytime sleepiness
Back Depression Inventory | From enrollment to the end of treatment at 12 weeks
  measures depression level min-max values: 0-63 Higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün Mesci, assoc prof, Study Director — Haydarpaşa Numune education and research Hospital
Locations (1):
- Haydarpaşa Numune Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol — https://haydarpasanumuneah.saglik.gov.tr/